CLINICAL TRIAL: NCT02186106
Title: The Effect of Oral Loading Doses of Cholecalciferol on the Serum Concentration of 25-OH-vitamin-D
Brief Title: Dosage Calculation for Vitamin D Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Rasmus Bo Jansen, MD, Bispebjerg Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-4-2011-094
Record Dates: First submitted 2014-07-03; First posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Deficiency, Vitamin D; Obesity
MeSH Terms: conditions — Vitamin D Deficiency; Obesity | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loading dose substitution (Experimental): Substituted with a highdose of cholecalciferol at study start
  Interventions: Drug: Cholecalciferol
- Historic controls (No Intervention): Control subjects from journal archive

INTERVENTIONS:
Drug: Cholecalciferol
  Other Names: Dekristol capsules of 20.000 IU pr. capsule
  Arms: Loading dose substitution

SUMMARY:
Severe vitamin D deficiency can be treated with oral loading doses of cholecalciferol. Our objective was to determine how to calculate the quantity of cholecalciferol needed for supplementation by single algorithm, usable on a patient-to-patient basis.

We've conducted two studies. Study 1 was done retroactively and included 88 patients treated for low vitamin D, 60 of those with a loading dose. The second study included 29 patients and aimed to test the validity of an algorithm based on data from study 1, which included patient BMI. Both studies used oral loading doses and daily supplementation of cholecalciferol.

ELIGIBILITY:
Inclusion Criteria:

* severe hypovitaminosis D (25OH-vit.D <25 nmol/L)

Exclusion Criteria:

* Malabsorption
* Renal disease
* Other treatment with vitamin D related products
* Patients with a recent travel history with suspected increased sun exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in baseline value of [25-OH-vitamin-D] | 1 week, 3 weeks and 3 months